CLINICAL TRIAL: NCT05649046
Title: Structuring of a Lung Cancer Screening Program Including Clinical, Radiological and Biological Phenotyping Useful for the Development of Individualized Risk Prediction Tools: PREVALUNG ETOILE
Acronym: PREVALUNG*
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RCAPHM22_0184; 2022-A01268-35 (Other: NUMERO IDRCB)
Record Dates: First submitted 2022-10-26; First posted 2022-12-13 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-02

CONDITIONS: Smoking-related Pathology; Atheroma; Chronic Bronchitis; Non-progressive Cancer > 5 Years; Lung Cancer
MeSH Terms: conditions — Plaque, Atherosclerotic; Bronchitis, Chronic; Lung Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients (Other)
  Interventions: Device: thoracic scan Low dose; Biological: BLOOD SAMPLE; Biological: FECES SAMPLE

INTERVENTIONS:
Device: thoracic scan Low dose — within 3 months after the V0 visit
Biological: BLOOD SAMPLE — within 3 months after the V0 visit
Biological: FECES SAMPLE — within 3 months after the V0 visit

SUMMARY:
Patients treated at the Hôpital Nord de Marseille for at least one smoking-related pathology (atheroma, chronic bronchitis, non-progressive cancer > 5 years) or with eligibility criteria for lung cancer screening (inclusion criteria in the NLST or NELSON studies or American recommendations) Interventional study with minimal risks and constraints, with evaluation of lung cancer prevalence; immunological, blood inflammatory and microbiota profile

Determine the maximum clinical, radiological, and biological phenotyping completeness rate following the implementation of a new lung cancer screening care pathway with multidimensional clinical, radiological, and biological phenotyping capabilities

ELIGIBILITY:
Inclusion Criteria:

Age 45- 75 years and

* Medical follow-up for a smoking-related pathology :
* atheroma
* chronic obstructive pulmonary disease / emphysema
* history of non evolving cancer > 5 years among: ENT, lung, breast, cervical, excreto-urinary cervix, excreto-urinary tract, bladder, esophagus, stomach, pancreas, liver, kidney, chronic myeloid leukemia chronic myeloid leukemia,
* daily smoking for at least 10 years prior to the disease Or

NLST inclusion criteria:

* Age 55 - 74 years
* Cumulative smoking ≥ 30 pack-years
* active or quit for less than 15 years Or

Inclusion criterion in NELSON:

* Age 50-75 years
* Smoking:
* > 15 cigarettes/D for more than 25 years or
* > 10 cigarettes /D for more than 30 years
* Active smoking or cessation < 10 years Or

New American recommendations :

* Age 50 - 80 years
* Smoking ≥20 PA
* Active or weaned <15 years

Exclusion Criteria:

history of cancer < 5 years (except carcinoma in situ of the uterine cervix, basal cell skin carcinoma basal cell carcinoma of the skin and prostate cancer with undetectable PSA)

* Symptoms of lung cancer (unintentional weight loss > 7 kg in 1 year, hemoptysis)
* known history of pulmonary nodule with specialized follow-up
* history of pulmonary fibrosis or pulmonary hypertension
* patient under guardianship or curatorship
* active pulmonary parenchymal infection
* severe cardiac or respiratory insufficiency (rest dyspnea)
* patient not affiliated to the social security system (beneficiary or beneficiary's right)
* Patient deprived of liberty
* Performance status (WHO) 2, 3 or 4
* Pregnant or breastfeeding women

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2023-01-23 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
number of complete phenotyping clinical, clinical | 18 months
number of complete phenotyping radiological | 18 months
number of complete phenotyping biological samples | 18 months

SECONDARY OUTCOMES:
Number of lung cancers diagnosed / Number of patients included | 18 MONTHS
Number of stage ≤ IIB lung cancers / number of lung cancers diagnosed | 18 MONTHS
Number of patients in partial smoking cessation / number of active smoking patients included | 18 MONTHS
Satisfaction assessment | 2 times (inclusion, 8 months)
  by scale SF-12
Assessment of ANXIETY | 2 times (inclusion, 8 months)
  by scale STAI-YA
Number of initial positive scans / number of initial scans | 18 months
Number of invasive procedures resulting in a diagnosis of a benign lesion / number of invasive procedures | 18 months
Number of cardiovascular events / number of patients included | 18 months
Number of oncological events (other than lung cancer) / number of patients included | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Emilie GARRIDO PRADALIE, Study Director — ASSIATANCE PUBLIQUE HOPITAUX DE MARSEILLE
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France